CLINICAL TRIAL: NCT05444374
Title: A Single-Arm, Multicenter, Phase II Study to Evaluate the Efficacy and Safety of Serplulimab Plus Bevacizumab in Combination With Chemotherapy in 1L Treatment of Patients With Untreated Recurrent or Metastatic Cervical Cancer
Brief Title: A Phase II Study of Serplulimab Plus Bevacizumab in Combination With Chemotherapy in 1L Treatment of Untreated Recurrent or Metastatic Cervical Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Guonan Zhang, Director, Head of Gynecologic Oncology Center, Sichuan Cancer Hospital and Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HLX10IIT05
Record Dates: First submitted 2022-06-29; First posted 2022-07-05 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Serplulimab plus Bevacizumab Combined With Chemotherapy (Experimental): Each cycle being 21 days, Cisplatin plus Paclitaxel up to 4-6 cycles, the maximum duration of treatment with Serplulimab is 2 years (up to 35 cycles).
  * Serplulimab, 300 mg IV, Day1 of each cycle
  * Bevacizumab, 7.5 mg/kg, IV, Day1 of each cycle
  * Cisplatin: 50 mg/m2, IV, Day1 of each cycle
  * Paclitaxel: 175 mg/m2, IV, Day1 of each cycle
  Interventions: Drug: Serplulimab; Drug: Bevacizumab

INTERVENTIONS:
Drug: Serplulimab — Recombinant anti-PD-1 humanized monoclonal antibody injection
Drug: Bevacizumab — Humanized anti-VEGF monoclonal antibody injection

SUMMARY:
This study is a single-arm, multicenter, Phase II study to evaluate the efficacy and safety of the treatment of Serplulimab plus Bevacizumab in combination with chemotherapy in 1L treatment of patients with untreated recurrent or metastatic cervical cancer.

Approximately 48 eligible subjects are planned to be enrolled across all sites.

The dosing regimen is: Serplulimab plus Bevacizumab combined with chemotherapy (cisplatin, paclitaxel).

Each cycle is 21 days (every 3 weeks). Subjects will receive Cisplatin plus Paclitaxel up to 4-6 cycles. The maximum duration of treatment with Serplulimab is 2 years (up to 35 cycles).

During the study treatment period, the subjects will receive imaging examination and response assessments every 6 weeks (± 7 days) in the first 48 weeks, every 9 weeks (± 7 days) in 48-96 weeks, and then every 12 weeks (± 7 days). After the treatment discontinuation visit, the subjects will enter the safety follow-up period and survival follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form (ICF)
2. Women, age ≥ 18 years and ≤ 75 years at time of signing ICF
3. Histologically or cytologically confirmed cervical cancer (pathological types: squamous cell carcinoma, adenocarcinoma [except mucinous adenocarcinoma], adenosquamous carcinoma)
4. Recurrent, progressive, or metastatic cervical cancer that is not amenable to surgery or radiotherapy/chemoradiotherapy (other than palliative radiotherapy to bone lesions). Recurrent and metastatic lesions should provide cytological and/or pathological biopsy evidence of cervical cancer metastasis as far as possible.
5. No systemic anti-tumor treatment for this recurrent, progressive or metastatic tumor. Note: a. Patients with initially diagnosed stage IVb disease should not have received systemic anti-tumor treatment; b. For patients previously treated with platinum-based first-line (neoadjuvant) adjuvant chemotherapy/radical chemoradiotherapy, the time from the last chemotherapy to disease recurrence is > 6 months; c. Patients treated with radiotherapy/concurrent chemoradiotherapy (only receiving platinum-based sensitization) can be enrolled after the completion of radiotherapy if they relapse outside the radiation field. If there is recurrence within the radiation field (RECIST 1.1 is met) and the target lesion is located in the radiation field, the patient can be enrolled more than 3 months after the completion of radiotherapy; d. For patients who have not received previous chemoradiotherapy, if chemoradiotherapy is required first (only platinum single agent sensitization is received), the patient can be enrolled more than 3 weeks after the completion of radiotherapy.
6. Prior anticancer TCM therapy must have ended ≥ 7 days prior to first study treatment (Cycle 1, Day 1) and all antineoplastic treatment-related AEs must have recovered to ≤ Grade 1 according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) 5.0 (except Grade 2 alopecia).
7. At least one measurable target lesion as assessed by the investigator per RECIST 1.1 within 4 weeks prior to enrollment.

   Note: Measurable target lesions should not have received local therapy such as radiotherapy (for lesions located in previously irradiated areas, target lesions can also be selected in case of definite progression [according to RECIST 1.1]).
8. ECOG PS score of 0 or 1 within 7 days prior to enrollment.
9. Expected survival ≥ 12 weeks.
10. Hepatitis B surface antigen (HBsAg) (-) and hepatitis B core antibody (HBcAb) (-). Hepatitis B virus deoxyribonucleic acid (HBV-DNA) < 2500 copies/mL or 500 IU/mL if HBsAg (+) or HBcAb (+).
11. Subjects who are HCV antibody (-) or HCV-RNA negative may be enrolled; if HCV-RNA is positive, subjects must have alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≤ 3 × ULN to be enrolled. Subjects with co-infection with hepatitis B and C are excluded (positive test for HBsAg or HBcAb and positive test for HCV antibody).
12. Adequate major organ function as defined by the following criteria (no transfusions, albumin, recombinant human thrombopoietin, or colony-stimulating factor [CSF] within 14 days prior to enrollment in this study):

Hematological system Neutrophils (ANC) 1.5 x 109/L Platelets (PLT) 100 x 109/L Hemoglobin (Hb) 90 g/L Hepatic function Total bilirubin (TB) ≤ 1.5 x upper limit of normal (ULN) Alanine aminotransferase (ALT) ≤ 2.5 × ULN;

* 5 × ULN for patients with liver metastases; Aspartate aminotransferase (AST) ≤ 2.5 × ULN;
* 5 × ULN for patients with liver metastases; Albumin ≥ 30 g/L Renal function Serum creatinine (Cr) ≤ 1.5 × ULN; Creatinine clearance ≥ 60 mL/min if > 1.5 × ULN (calculated according to Cockcroft-Gault formula) Coagulation function Activated partial thromboplastin time (APTT) ≤ 1.5 x ULN Prothrombin time (PT) or international normalized ratio (INR) ≤ 1.5 x ULN 13. Female patients must meet: i. Menopause (defined as no menses for at least 1 year and no other confirmed cause other than menopause), or ii. Have been surgically sterilized (removal of ovaries and/or uterus), or iii. Childbearing potential, but must meet:

  * Must have a negative serum pregnancy test within 7 days prior to randomization, and
  * Agree to practice contraception with an annual failure rate of < 1% or remain abstinent (refrain from heterosexual intercourse) (from signing the ICF to at least 6 months after the last dose of investigational drug and at least 6 months after the last dose of chemotherapeutic drugs) (methods of contraception with an annual failure rate of < 1% include bilateral tubal ligation, male sterilization, correct use of hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper-containing intrauterine devices or condoms), AND
  * Do not breastfeed.

Exclusion Criteria:

Patients who meet any of the following exclusion criteria will not be enrolled in the study:

1. Other active malignancy within 2 years or concurrently. Cured localized tumors, such as cutaneous basal cell carcinoma, cutaneous squamous cell carcinoma, superficial bladder cancer and breast carcinoma in situ, can be enrolled.
2. Patients who are scheduled for or have received prior organ or bone marrow transplantation.
3. Patients with uncontrolled pleural effusion, pericardial effusion or ascites.
4. Central nervous system (CNS) or leptomeningeal metastases confirmed by imaging studies or pathology.
5. Myocardial infarction within 6 months prior to enrollment, poorly controlled arrhythmia (including QTc interval ≥ 470 ms for females) (QTc interval calculated using Fridericia's formula).
6. Class III-IV cardiac dysfunction according to New York Heart Association (NYHA) criteria or echocardiography: left ventricular ejection fraction (LVEF) < 50%.
7. Poorly controlled hypertension (defined as systolic blood pressure ≥ 150 mmHg and/or diastolic blood pressure ≥ 100 mmHg), previous hypertensive crisis or hypertensive encephalopathy.
8. Human immunodeficiency virus (HIV) infection.
9. Patients with active pulmonary tuberculosis.
10. Patients with previous and current interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonitis, severely impaired pulmonary function, etc., which may interfere with the detection and management of suspected drug-related pulmonary toxicity.
11. Patient has known active or suspected autoimmune disease. Patients with immune-related hypothyroidism on thyroid hormone replacement therapy and patients with well-controlled type I diabetes are allowed. Recovered Vitiligo or childhood asthma/allergies that do not require intervention or that do not require any intervention in adulthood are allowed.
12. Treatment with a live vaccine within 28 days prior to enrollment. However, inactivated viral vaccines for seasonal influenza are allowed, but live attenuated influenza vaccines for intranasal use are not allowed.
13. Patients requiring systemic corticosteroids (> 10 mg/day prednisone efficacy dose) or other immunosuppressive medications within 14 days prior to enrollment or during the study. However, patients were permitted to use topical or inhaled corticosteroids and adrenal glucocorticoid replacement at doses ≤ 10 mg/day prednisone for efficacy in the absence of active autoimmune disease.
14. Any active infection requiring systemic anti-infective therapy within 14 days prior to enrollment.
15. Major surgery within 28 days prior to enrollment, this study Major surgery is defined as surgery that requires at least 3 weeks of recovery from surgery to be able to receive treatment for this study. Patients with tumor aspirate or lymph node harvest biopsy were allowed to enroll.
16. The patient has previously received other antibodies/drugs against immune checkpoints, such as PD-1, PD-L1, cytotoxic T lymphocyte-associated antigen 4 (CTLA-4) and other treatments.
17. Ongoing participation in another clinical study, or planned initiation of treatment in this study less than 14 days from the end of treatment in the previous clinical study.
18. Presence of free air in the abdomen that cannot be explained by puncture or recent surgical procedure.
19. Presence of bladder or rectal fistula at screening.
20. Acute intestinal obstruction or incomplete obstruction within 6 months. However, patients with complete response (CR) after surgical treatment may be enrolled.
21. Uncontrolled tumor-related pain.
22. Known history of serious allergy to any monoclonal antibody.
23. Known hypersensitivity to any of the cisplatin or paclitaxel components.
24. Pregnant or lactating women.
25. Patient has a known history of psychiatric drug abuse or drug abuse; patient has a history of alcohol abuse.
26. The patient has other factors that, in the judgment of the investigator, may lead to forced early termination of the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 2 years
  Defined as the proportion of patients whose best overall response is a partial response (PR) or a CR during the study, as determined by investigators

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Up to approximately 2 years
  Defined as the time from enrollment to the first occurrence of disease progression or death from any cause, whichever occurs first, as determined by investigators
Duration of Response (DOR) | Up to approximately 2 years
  Defined as the time from the first occurrence of a documented objective response (CR or PR) to disease progression, or death from any cause, whichever occurs first
Disease Control Rate (DCR) | Up to approximately 2 years
  Percentage of Participants Achieving Complete Response (CR) and Partial Response (PR) and Stable Disease (SD)
3-year Overall Survival (OS) | Up to approximately 2 years
  Defined as the time from enrollment to death, regardless of cause of death. For subjects who had not been reported to have died at the time of analysis, the date they were last known to be alive was used as the censoring date for OS
Number of Participants Who Experience One or More Adverse Events (AEs) | From randomization through 30 days after last dose of study treatment (Up to approximately 25 months)
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Guonan Zhang, Principal Investigator — Sichuan Cancer Hospital and Research Institute
Locations (4):
- China (4):
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Sicchuan Cancer Hospital, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Waggoner SE. Cervical cancer. Lancet. 2003 Jun 28;361(9376):2217-25. doi: 10.1016/S0140-6736(03)13778-6. PMID 12842378
- [Background] Pfaendler KS, Tewari KS. Changing paradigms in the systemic treatment of advanced cervical cancer. Am J Obstet Gynecol. 2016 Jan;214(1):22-30. doi: 10.1016/j.ajog.2015.07.022. Epub 2015 Jul 26. PMID 26212178
- [Background] Todo Y, Watari H. Concurrent chemoradiotherapy for cervical cancer: background including evidence-based data, pitfalls of the data, limitation of treatment in certain groups. Chin J Cancer Res. 2016 Apr;28(2):221-7. doi: 10.21147/j.issn.1000-9604.2016.02.10. PMID 27199520
- [Background] Verma J, Monk BJ, Wolfson AH. New Strategies for Multimodality Therapy in Treating Locally Advanced Cervix Cancer. Semin Radiat Oncol. 2016 Oct;26(4):344-8. doi: 10.1016/j.semradonc.2016.05.003. Epub 2016 May 26. PMID 27619255
- [Background] Moore DH, Blessing JA, McQuellon RP, Thaler HT, Cella D, Benda J, Miller DS, Olt G, King S, Boggess JF, Rocereto TF. Phase III study of cisplatin with or without paclitaxel in stage IVB, recurrent, or persistent squamous cell carcinoma of the cervix: a gynecologic oncology group study. J Clin Oncol. 2004 Aug 1;22(15):3113-9. doi: 10.1200/JCO.2004.04.170. PMID 15284262